CLINICAL TRIAL: NCT00345553
Title: Biliary Atresia Study in Infants and Children (BASIC)
Brief Title: Biliary Atresia Study in Infants and Children
Acronym: BASIC
Status: Recruiting | Type: Observational
Sponsor: Arbor Research Collaborative for Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: BASIC Study - ChiLDReN Network; U01DK103149 (NIH); U01DK103140 (NIH); U01DK103135 (NIH); U01DK084575 (NIH); U01DK084538 (NIH); U01DK084536 (NIH); U01DK062503 (NIH); U01DK062500 (NIH); U01DK062497 (NIH); U01DK062481 (NIH); U01DK062470 (NIH); U01DK062466 (NIH); U01DK062456 (NIH); U01DK062453 (NIH); U01DK062452 (NIH); U01DK062445 (NIH); U01DK062436 (NIH); U24DK062456 (NIH)
Record Dates: First submitted 2006-06-27; First posted 2006-06-28 (Estimated); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Biliary Atresia
Keywords: Biliary Atresia; Cholestasis
MeSH Terms: conditions — Biliary Atresia; Cholestasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples of blood will be collected for research purposes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 1: Biliary atresia subjects who have their native liver

SUMMARY:
Little is known about the factors that cause biliary atresia nor the factors that influence disease progression. The purpose of this study is to collect the pertinent clinical information, genetic material and body fluid samples to enable investigators to address the following aims: To identify the gene or genes implicated in the etiology of BA; To characterize the natural history of the older, non-transplanted child with BA.

DETAILED DESCRIPTION:
Little is known about the factors that cause biliary atresia nor the factors that influence disease progression. A variety of genetic, autoimmune and environmental influences have been hypothesized to be important. Most studies to date have focused on the neonate and young child with BA, yet the older surviving child with BA can provide important information about genetics, as well as, natural history.

The purpose of this study is to collect the pertinent clinical information, genetic material and body fluid samples to enable investigators to address the following hypotheses:

Hypothesis 1: A genetic defect is a likely causative factor for BA among children with BA and multiple congenital anomalies.

Hypothesis 2a: Sentinel events such as variceal bleeding, ascites and growth failure are earlier predictors of death or need for liver transplantation than the pediatric end-stage liver disease score (PELD).

Hypothesis 2b: Health related quality of life will be impaired compared to healthy age matched children and relate to severity of illness.

Hypothesis 2c: Growth failure as measured by anthropometrics and nutritional supplementation will be predictive of onset of sentinel events (ascites, variceal bleed, death, and transplant) in the following 24 months.

This study will be performed by the Childhood Liver Disease Research Network (ChiLDReN), a National Institute of Diabetes & Digestive and Kidney Diseases (NIDDK) funded network.

ELIGIBILITY:
Inclusion Criteria:

1. Participants need to have a confirmed diagnosis of BA determined by chart review including review of pertinent diagnostic biopsy reports, radiologic reports and surgical reports (if surgery was performed).
2. Participants need to be >6 months of age up to and equal to the age of 20 (participants enrolled at 20 years of age will have one visit).
3. Participants with their native liver.
4. Parent, guardian or participant (if 18 years of age or older) is willing to provide informed consent and, when appropriate, the participant is willing to assent.

Exclusion Criteria:

1. Currently participating in the ChiLDReN study PROBE.
2. Inability to confirm original diagnostic evaluation of biliary atresia.
3. Inability or unwillingness of family or participant to participate in all scheduled visits.
4. History of liver transplantation.

Ages: 6 Months to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Recruitment will be open to any eligible subject. The method of contacting the study subjects will conform to local IRB guidelines, but in general: the parents or guardians of all eligible subjects at each ChiLDReN center, or the subjects themselves if 18 years of age or older, will be approached to participate. New patients who are not participating in ChiLDReN study PROBE may be approached for study participation, but will not be eligible for enrollment until 6 months of age.
Sampling Method: Non-Probability Sample
Enrollment: 1265 (Estimated)
Dates: Start 2006-05-16 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
To identify the gene or genes implicated in the etiology of BA | Specimens for this aim are collected once during study, usually at baseline.
  The genetics of BA may be investigated on two levels. The first is to identify a group of patients whose etiology is a result of a genetic defect and the second is to examine the influence of genetics on disease acquisition.

SECONDARY OUTCOMES:
Define the natural history of the older, non-transplanted child with biliary atresia | Observational information collected at entrance into study as well as at each yearly follow-up visit.
  Understanding the natural history of a disease is a prerequisite to interpreting disease severity, identifying patterns of illness, identifying early predictors of outcome and understanding the advantages or trade-offs of therapeutic interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjiv Harpavat, MD, Study Chair — Texas Children's/Baylor College of Medicine; Ed Doo, MD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK); John C Magee, MD, Principal Investigator — University of Michigan; Lisa Henn, PhD, Principal Investigator — Arbor Research Collaborative for Health - Data Coordinating Center; Katrina Loh, MD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (16):
- United States (15):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of California at San Francisco, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta - Emory University, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Children's Hospital, Indianapolis, Indiana
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Mount Sinai Medical Center, New York, New York
  - Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Texas Children's Hospital (Baylor College of Medicine), Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The data will be transferred to NIDDK at the end of the study.

REFERENCES:
- [Derived] Ng VL, Haber BH, Magee JC, Miethke A, Murray KF, Michail S, Karpen SJ, Kerkar N, Molleston JP, Romero R, Rosenthal P, Schwarz KB, Shneider BL, Turmelle YP, Alonso EM, Sherker AH, Sokol RJ; Childhood Liver Disease Research and Education Network (CHiLDREN). Medical status of 219 children with biliary atresia surviving long-term with their native livers: results from a North American multicenter consortium. J Pediatr. 2014 Sep;165(3):539-546.e2. doi: 10.1016/j.jpeds.2014.05.038. Epub 2014 Jul 9. PMID 25015575
- See also: Childhood Liver Disease Research Network (ChiLDReN) website — http://www.childrennetwork.org